CLINICAL TRIAL: NCT02502045
Title: A Study to Examine the Effect of Therapeutic Light on Sleep, Circadian Rhythm, and Global Function in Women With Alzheimer's Disease
Brief Title: Effect of Therapeutic Light on Sleep, Circadian Rhythm, and Global Function in Women With Alzheimer's
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1310012895
Record Dates: First submitted 2015-07-16; First posted 2015-07-17 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning Simulated Sunlight (Experimental): Timed morning simulated sunlight (Philips Wake Up Light, Model HF3520) peaking at 300 lux delivered over a 40 minute ramp between 5-9 a.m. for 14 consecutive days. A flexible window of has been allowed to accommodate participants and care routines.
  Interventions: Device: Morning Simulated Sunlight
- Non-Therapeutic Red Light (Placebo Comparator): Non-therapeutic red light control at 5 lux will be used as the control condition
  Interventions: Device: Non-therapeutic Red Light

INTERVENTIONS:
Device: Morning Simulated Sunlight — Timed morning simulated sunlight (Philips Wake Up Light, Model HF3520) peaking at 300 lux delivered over a 40 minute ramp between 5-9 a.m. for 14 consecutive days
  Arms: Morning Simulated Sunlight
Device: Non-therapeutic Red Light — Non-therapeutic red light control at 5 lux will be used as the control condition
  Arms: Non-Therapeutic Red Light

SUMMARY:
Determine effect and duration of effect of timed therapeutic light compared to control light on parameters of circadian rhythmicity, physiologic plasticity, sleep, and global function in women with Alzheimer's Disease.

DETAILED DESCRIPTION:
The impact of disturbed sleep on cognition and functional domains is vitally important to study in order to increase our understanding of Alzheimer's disease (AD) phenomenology. Research has shown that the severity of sleep disturbance and dementia advance in parallel and possibly in a manner amenable to therapeutic intervention. In AD, sleep disruption is characterized by changes in sleep architecture. It is our contention that neuropathology specific to AD alters the circadian system at the suprachiasmatic nucleus (SCN). Environmental light is the most powerful regulator of this circadian system,4,5 and is known to have a significant regulatory effect on pineal melatonin synthesis and secretion via the SCN and multisynaptic pathways downstream from the SCN. This study will explore further the efficacy of a particular type of therapeutic light intervention in regulating the circadian system in AD, using data analytic methods capable of detecting changes at multiple time scales. Our central hypothesis is that properly-timed light exposure in individuals with AD will synchronize disorganized circadian and sleep-wake rhythms and improve functional plasticity [approximate entropy (ApEn), fractal dimension (FD)], thereby resulting in increased sleep efficiency (SE), reductions in sleep fragmentation (SF), reduced excessive daytime sleepiness (EDS) and dementia-related behaviors, and improvements in cognition and other daytime behaviors. Women are nearly twice as likely as men to develop AD due to longer life expectance and emerging evidence. In light of this increased risk and also to enhance other aspects of biological uniformity in our study, this project will investigate women with AD.

ELIGIBILITY:
Inclusion Criteria:

1. baseline sleep efficiency index < .85
2. Mini-Mental State Exam-2 Standard Version (MMSE-2:SV) score of 0-20
3. be medically stable

Exclusion Criteria:

1. received light treatment in last 3 months
2. are totally blind in both eyes, have photosensitivity or photophobia, Parkinsons disease, known untreated sleep apnea or other sleep disorders, seizure disorder, bipolar, schizophrenia, are actively receiving chemotherapy or radiation therapy for cancer.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in sleep characteristics | 2 weeks
  Change in sleep characteristics and rest-activity rhythm after 2 weeks of light therapy as measured by actigraphy

CONTACTS AND LOCATIONS:
Overall Officials: LuAnn Etcher, PhD, Principal Investigator — Yale University
Locations (1):
- Botsford Continuing Care, Farmington Hills, Michigan, United States